CLINICAL TRIAL: NCT00624767
Title: A Phase 2, Randomized, Crossover Study to Evaluate the Effect of Intranasal Insulin and NovoLog on Postprandial Glycemic Control in Type 2 Diabetic Patients
Brief Title: A Study to Evaluate the Effect of Nasal Insulin on Postprandial Glycemic Control in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nastech Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sherwyn Schwartz, MD, Diabetes and Glandular Disease Research Associates
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C08-002
Record Dates: First submitted 2008-02-07; First posted 2008-02-27 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus
Keywords: insulin; insulin aspart; Type 2 Diabetes; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Insulin Nasal Spray
  Interventions: Drug: Insulin (recombinant human insulin)
- 2 (Active Comparator): NovoLog
  Interventions: Drug: NovoLog

INTERVENTIONS:
Drug: Insulin (recombinant human insulin) — Insulin Nasal Spray at doses up to 200 IU.
  Other Names: recombinant human insulin
  Arms: 1
Drug: NovoLog — NovoLog at doses up to 30 IU
  Other Names: insulin aspart
  Arms: 2

SUMMARY:
Insulin is a hormone which is produced by the human pancreas for the lowering of blood sugar. In patients who don't produce enough insulin, additional insulin must be given several times per day by injections. Nastech Pharmaceutical Company Inc. has developed a new insulin nasal spray, as a possible way to improve patient compliance with intensive insulin treatment plans. This study is being conducted to see how Nastech's insulin nasal spray affects post-meal glucose levels compared with rapid acting insulin (i.e., insulin aspart) in Type 2 diabetics who are already taking oral antidiabetic medications and/or insulin therapy. Insulin aspart is marketed as NovoLog® in the United States. The safety of insulin nasal spray and how well it is tolerated as compared to NovoLog will also be evaluated.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the effect on postprandial glucose levels and safety of Nastech's insulin nasal spray compared with a rapid acting insulin (i.e., insulin aspart) in Type 2 diabetics. Insulin aspart is marketed as NovoLog® in the United States and NovoRapid® in Europe.

The target for the patient titration scheme is that the 60 minute glucose reading does not increase more than 3.3 mmol/L (60 mg/dL) above the fasting glucose level AND does not result in hypoglycemia at any time within four hours post meal.

NovoLog doses will be chosen based on a patient's current prandial insulin dose, or a dose of 25% of their basal insulin dose or 8 IU if on oral antidiabetic therapy only. Then patients will be titrated up or down for up to three additional consecutive treatments from the initial dose (potential of 4 doses of NovoLog). Once a patient reaches their target titrated dose with NovoLog they are then titrated with nasal insulin.

The nasal doses will correspond to the injectable dose based on bioavailability. For example, the nasal formulation being tested in this study has a 17%-28% bioavailability compared to NovoLog. Therefore a 25 IU nasal dose corresponds to a 4-7 IU NovoLog injectable dose. The patients will be titrated up or down per dose with nasal insulin for up to three additional consecutive treatments from the initial dose (potential of 4 doses of nasal insulin). Once a patient has been successfully titrated with NovoLog and then nasal insulin, they will be randomized to a two-way crossover where they will be given NovoLog and Nasal insulin. There will be at least a 20 hour washout period between titration and randomization stages. Patients will be monitored for symptoms consistent with hypoglycemia. If needed, treatment with oral carbohydrates such as glucose tablets, fruit juices, non-diet soda will be provided. In the event a patient is unable to take oral glucose, intravenous 20% glucose solution (D20) will be available.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months
* Type 2 diabetics on oral antidiabetic medicines and/or insulin therapies

Exclusion Criteria:

* Patients taking intermediate acting insulin such as NPH
* Recurrent severe hypoglycemia
* Patients with late diabetic complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect on postprandial glycemic control of intranasal insulin compared to NovoLog | 4 hour Profile

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of intranasal insulin compared to NovoLog | 4 hour Profile

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, MD, Principal Investigator — Diabetes and Glandular Disease Research Associates
Locations (1):
- Diabetes and Glandular Disease Research Associates, San Antonio, Texas, United States